CLINICAL TRIAL: NCT02047864
Title: Long-term Effects of Creatine Supplementation and Exercise Training on Bone Mineral Density and Bone Strength in Postmenopausal Women
Brief Title: Effect of Creatine Supplementation and Exercise on Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 300561
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Osteoporosis; Sarcopenia
Keywords: Osteoporosis; Sarcopenia; Strength; Bone; Muscle; Creatine
MeSH Terms: conditions — Osteoporosis; Sarcopenia | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Creatine monohydrate (Experimental): Creatine monohydrate to be given during a resistance training program
  Interventions: Dietary Supplement: Creatine monohydrate
- Sugar pill (Placebo Comparator): Placebo to be given during a resistance training program
  Interventions: Dietary Supplement: Creatine monohydrate

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate

SUMMARY:
Osteoporosis is an important health problem, costing the Canadian health care system over $2 billion per year. Loss of bone mineral and bone fragility is especially prevalent in postmenopausal women. Of all osteoporotic fractures, hip fractures are the most traumatic. Creatine monohydrate is a nutritional supplement that is often combined with strength training to increase strength and muscle mass. The investigators recently completed a pilot study in a small number of postmenopausal women (n=33) that showed that creatine monohydrate significantly improved hip bone mineral density during a 1-year resistance training program. In our current proposal the investigators want to determine whether creatine combined with strength training can have an even larger effect on bone mineral density at the hip if given over 2 years in a large group of postmenopausal women (n=240). The investigators also want to determine whether this leads to reduced fractures in these women for up to a year after completing the creatine and strength training program.

DETAILED DESCRIPTION:
Age-related bone and muscle loss is a major risk factor for falls, injuries, and fracture and, as Canada's population is aging, prevalence of such health concerns is escalating. Osteoporosis alone is estimated to cost the Canadian health care system $2.3 billion per year or 1.3%, of Canada's total healthcare budget. Postmenopausal women are at high risk of osteoporosis and experience the highest rate of hip fracture, resulting in disability, loss of physical function and premature death. The investigators' study aims to improve bone mass and bone strength at the most clinically relevant bone site, the femoral neck, in order to reduce the risk of hip fracture. Specifically, it will determine the effects of a nutritional supplement (creatine monohydrate) combined with exercise training on bone mineral density (BMD) at the proximal femur in postmenopausal women. .

Creatine monohydrate is found in small amounts in meats and fish and, when taken as a nutritional supplement, increases muscle mass and strength. The investigators have conducted a number of preliminary studies showing that when a creatine supplement is taken during a resistance training program, urinary markers of bone resorption (i.e. bone catabolism) are reduced compared to placebo. The investigators recently completed a small 12-month randomized controlled trial in 33 postmenopausal women who either supplemented with creatine monohydrate (10 g/d) or placebo during a resistance training program. Bone mineral density of the femoral neck decreased by 0.5% in the creatine group, and 3.9% in the placebo group (p<0.05 between groups). This proposed randomized controlled trial will replicate the investigators' pilot design for longer duration (i.e. 2 years) to determine if sustained supplementation with creatine monohydrate combined with exercise training can induce a clinically significant difference in bone mineral density at the femoral neck (the investigators estimate a 5% difference between creatine and placebo groups capable of predicting a significant reduction in fracture risk).

This trial will use a randomized, double blind, placebo controlled, parallel group, repeated measures design, performed at the Universities of Saskatchewan and Regina. Post-menopausal women (n=240) will be randomized to creatine (10g/d) or placebo groups while participating in an exercise program (resistance training and walking) three times per week for 24 months. The investigators' main dependent variable is femoral neck bone mineral density, which will be assessed at baseline, 12, and 24 months. Secondary variables to be assessed at the same time points include geometric properties of the proximal femur (predictors of bone strength), lumbar spine bone mineral density, ultrasound measurements of bone at the distal radius and tibia (predictive of the architectural integrity of bone), lean tissue mass, muscular strength, dynamic balance, and gait speed. The investigators will assess incidence of falls and fractures at the same time points and also at 12 months post-intervention (i.e. at 36 months). The results of this study have clinical potential, providing physicians and health-care professionals evidence-based advice to give to postmenopausal women interested in taking creatine as a novel strategy to increase bone mineral density and prevent osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Low or moderate risk of fracture

Exclusion Criteria:

* High risk of fracture
* Have taken any bone-altering drugs within the previous 12 months
* Have taken creatine monohydrate in the previous 12 months
* Currently taking systemic corticosteroids
* Have Crohn's Disease or Cushings Disease
* Have severe osteoarthritis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in femoral neck bone mineral density | baseline, 12 months, 24 months

SECONDARY OUTCOMES:
Change from baseline in total hip bone mineral density | baseline, 12 months, 24 month
Change from baseline in trochanter bone mineral density | baseline, 12 months, 24 month
Change from baseline in Wards bone mineral density | baseline, 12 months, 24 months
Change from baseline in lumbar spine bone mineral density | baseline, 12 months, 24 months
Change from baseline in whole body bone mineral density | baseline, 12 months, 24 months
Change from baseline in hip geometric properties | baseline, 12 months, 24 months
  The geometric properties include cross-sectional area, subperiosteal width, cross-sectional moment of inertia, and section modulus at the femoral neck, intertrochanteric site, and the femoral shaft
Change in radius speed of sound | baseline, 12 months, 24 months
Change from baseline in tibial speed of sound | Baseline, 12 months, 24 months
Change from baseline in lean tissue mass | baseline, 12 months, 24 months
Change from baseline in squat maximal strength | baseline, 12 months, 24 months
Change from baseline for chest press strength | baseline, 12 months, 24 months
Change from baseline for dynamic balance | Baseline, 12 months, 24 months
Change from baseline for walking speed | Baseline, 12 months, 24 months
Number of falls | 12, 24, and 36 months
Number of fractures | 12, 24, and 36 months
Changes from baseline in blood markers of liver and kidney function and complete blood cell count | baseline, 12 months, 24 months
Changes in diet from baseline | Baseline, 12 months, 24 months
Changes in physical activity from baseline | Baseline, 12 months, 24 months
Changes from baseline in adverse events | Baseline, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, PhD, Principal Investigator — University of Saskatchewan; Darren Candow, PhD, Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - University of Regina, Regina, Saskatchewan
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chilibeck PD, Candow DG, Gordon JJ, Duff WRD, Mason R, Shaw K, Taylor-Gjevre R, Nair B, Zello GA. A 2-yr Randomized Controlled Trial on Creatine Supplementation during Exercise for Postmenopausal Bone Health. Med Sci Sports Exerc. 2023 Oct 1;55(10):1750-1760. doi: 10.1249/MSS.0000000000003202. Epub 2023 May 5. PMID 37144634